CLINICAL TRIAL: NCT00179634
Title: Using Visual Milieu Enrichment and Guided Visualization to Augment Patient Well-being and Post-surgical Recovery
Brief Title: Study of Fine Art Photographs and Visualization Tapes to Improve Surgical Recovery in Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expired for lack of continuing review
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, James Rodrigue, Professor of Psychology in the Department of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004P000115; West
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Breast Neoplasms
Keywords: Mastectomy; Randomized Controlled Trial; Imagery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Usual Care
- 2 (Experimental): Usual care and exposure to a visually enriched milieu (landscape photograph)
  Interventions: Behavioral: Visual Milieu Enhancement (Fine art photograph)
- 3 (Experimental): Usual care, exposure to a visually enriched milieu and audio taped guided visualization with healing suggestions.
  Interventions: Behavioral: Visualization relaxation; Behavioral: Visual Milieu Enhancement (Fine art photograph)

INTERVENTIONS:
Behavioral: Visualization relaxation
  Arms: 3
Behavioral: Visual Milieu Enhancement (Fine art photograph)
  Arms: 2; 3

SUMMARY:
This is a study to assess whether healing suggestions and enhancing visual milieu (large fine art photographs) will improve mental and physical measures of well-being and recovery from surgery. The study will compare breast cancer patients undergoing identical skin sparing mastectomy and reconstruction surgery randomized to three groups:

1. Usual care control group
2. Usual care and exposure to fine art photograph
3. Usual care and fine art photograph and guided visualization tapes.

DETAILED DESCRIPTION:
In the course of surgical procedures and hospitalization, patients are stressed not only by the discomforts and anxieties associated with their illness and treatment but also by the sterile, intimidating medical environment, with no access to the natural environment. Clinical studies from environmental medicine have suggested that during hospital confinement patients benefit from visually pleasing décor. Enhancing the medical milieu can alleviate patient anxiety and discomfort as well as improve markers of stress such as blood pressure and requirement for analgesics. In addition, research has shown the effectiveness of stress reduction approaches such as Relaxation Response, Guided Imagery, and Hypnosis in mediating clinical psychophysiology overall. Such studies have also shown the lowering of stress levels, inducing faster recovery from surgical anesthesia and perhaps even speeding physical healing overall. Use of these techniques has been shown to give people a greater sense of self-control as well and reduce stress reactions that affect health.

The proposed study represents the next step testing clinical efficacy of a behavioral medicine intervention with breast cancer patients undergoing mastectomy and reconstruction surgery. The current study extends prior research on accelerating healing outcomes through the use of non-pharmacological mental interventions. One prior study demonstrated accelerated bone fracture healing using hypnosis in otherwise healthy young adults. A second study showed enhanced post-surgical wound healing in healthy women undergoing reduction mammoplasty. The current study will generate new data about enhancing outcomes for breast cancer patients undergoing mastectomy and reconstruction. The goal of the trial is to determine whether these ancillary treatments enhance psychological and physical post-surgical recovery as compared to usual care only. The study provides an upside potential to enhance patient well being and to accelerate post-surgical recovery with minimal risk. Should significant positive findings result from this study, it will constitute a pilot test of such modifications of the healthcare delivery environment with an eye toward stimulating greater patient well being and shorter length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage 0, I, or II breast cancer
* Skin sparing mastectomy with transverse rectus abdominal muscle (TRAM) or deep inferior epigastric perforator (DIEP) flap reconstruction planned
* Ability to give informed consent
* Working knowledge of English

Exclusion Criteria:

* Physical inability to comply to study protocol
* Diabetes
* Current smokers
* Acute psychosis
* Mental retardation
* Language barriers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03-27 (Actual); Study Completion 2008-03-27 (Actual)

PRIMARY OUTCOMES:
Mood disturbance (Profile of Mood States short form) | 4 weeks
Post-operative pain | 4 weeks
Presence of skin necrosis | 4 weeks
Presence of hematoma | 4 weeks
Presence of infection | 4 weeks
Length of hospital stay | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Troyan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hartig T, Evans GW, Jammer LD, Davis DS, Garling T. Tracking restoration in natural and urban field settings. Journal of Environmental Psychology 23:109-23, 2003
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899
- [Background] Lembo T, Fitzgerald L, Matin K, Woo K, Mayer EA, Naliboff BD. Audio and visual stimulation reduces patient discomfort during screening flexible sigmoidoscopy. Am J Gastroenterol. 1998 Jul;93(7):1113-6. doi: 10.1111/j.1572-0241.1998.00339.x. PMID 9672340
- [Background] Tusek DL, Church JM, Strong SA, Grass JA, Fazio VW. Guided imagery: a significant advance in the care of patients undergoing elective colorectal surgery. Dis Colon Rectum. 1997 Feb;40(2):172-8. doi: 10.1007/BF02054983. PMID 9075752
- [Background] Blankfield RP. Suggestion, relaxation, and hypnosis as adjuncts in the care of surgery patients: a review of the literature. Am J Clin Hypn. 1991 Jan;33(3):172-86. doi: 10.1080/00029157.1991.10402927. PMID 2012007
- [Background] Benson H, Friedman R. Harnessing the power of the placebo effect and renaming it "remembered wellness". Annu Rev Med. 1996;47:193-9. doi: 10.1146/annurev.med.47.1.193. PMID 8712773
- [Background] Ewin DM.The effect of hypnosis and mental set on major surgery and burns. Psychiatric Annals 16:115-118, 1986.
- [Background] Halpin LS, Speir AM, CapoBianco P, Barnett SD. Guided imagery in cardiac surgery. Outcomes Manag. 2002 Jul-Sep;6(3):132-7. PMID 12134377
- [Background] Hoffman JW, Benson H, Arns PA, Stainbrook GL, Landsberg GL, Young JB, Gill A. Reduced sympathetic nervous system responsivity associated with the relaxation response. Science. 1982 Jan 8;215(4529):190-2. doi: 10.1126/science.7031901.
- [Background] Holden-Lund C. Effects of relaxation with guided imagery on surgical stress and wound healing. Res Nurs Health. 1988 Aug;11(4):235-44. doi: 10.1002/nur.4770110405. PMID 3043570
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Background] Glaser R, Kiecolt-Glaser JK, Marucha PT, MacCallum RC, Laskowski BF, Malarkey WB. Stress-related changes in proinflammatory cytokine production in wounds. Arch Gen Psychiatry. 1999 May;56(5):450-6. doi: 10.1001/archpsyc.56.5.450. PMID 10232300
- [Background] Ginandes CS, Rosenthal DI. Using hypnosis to accelerate the healing of bone fractures: a randomized controlled pilot study. Altern Ther Health Med. 1999 Mar;5(2):67-75. PMID 10069091
- [Background] Ginandes C, Brooks P, Sando W, Jones C, Aker J. Can medical hypnosis accelerate post-surgical wound healing? Results of a clinical trial. Am J Clin Hypn. 2003 Apr;45(4):333-51. doi: 10.1080/00029157.2003.10403546. PMID 12722936